CLINICAL TRIAL: NCT01001494
Title: Efficacy and Safety of Aclidinium Bromide at Two Dose Levels vs Placebo When Administered to Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Aclidinium Bromide at Two Dose Levels Versus Placebo Administered in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/34; ATTAIN
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; antimuscarinic; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aclidinium bromide 200 μg bid (Experimental): Aclidinium bromide 200 μg twice-daily via inhalation
  Interventions: Drug: Aclidinium bromide 200 μg bid
- Aclidininum bromide 400 μg bid (Experimental): Aclidinium bromide 400 μg twice-daily via inhalation
  Interventions: Drug: Aclidinium bromide 400 μg bid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide 200 μg bid — Aclidinium bromide 200 μg twice-daily via inhalation by the Eklira Genuair® inhaler: 1 puff in the morning and evening for 24 weeks
  Arms: Aclidinium bromide 200 μg bid
Drug: Aclidinium bromide 400 μg bid — Aclidinium bromide 400 μg twice-daily via inhalation by the Eklira Genuair® inhaler: 1 puff in the morning and evening for 24 weeks
  Arms: Aclidininum bromide 400 μg bid
Drug: Placebo — Placebo twice-daily by inhalation for 24 weeks
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the long term bronchodilator efficacy, safety and tolerability of inhaled aclidinium bromide at two dose levels compared to placebo in COPD patients and the benefits of the product in disease-related health status, COPD symptoms and COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients aged ≥40 with stable moderate to severe COPD (GOLD guidelines).
* Post-salbutamol (FEV1) < 80% and ≥30% of predicted normal value and Post-salbutamol FEV1/FVC < 70%.
* Current or ex-smokers of ≥10 pack-years.

Exclusion Criteria:

* Patients with no history or current diagnosis of asthma.
* No evidence of an exacerbation within 6 weeks prior to the screening visit.
* No evidence of clinically significant respiratory and/or cardiovascular conditions or laboratory abnormalities.
* No contraindication to use of anticholinergic drugs such as known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (106):
- Czechia (10):
  - Almirall Investigational Sites#4, Benešov
  - Almirall Investigational Sites#9, Jaroměř
  - Almirall Investigational Sites#3, Liberec
  - Almirall Investigational Sites#2, Lovosice
  - Almirall Investigational Sites#1, Neratovice
  - Almirall Investigational Sites#11, Prague
  - Almirall Investigational Sites#6, Prague
  - Almirall Investigational Sites#12, Prague
  - Almirall Investigational Sites#7, Prague
  - Almirall Investigational Sites#10, Strakonice
- France (5):
  - Almirall Investigational Sites#3, Clermont-Ferrand
  - Almirall Investigational Sites#2, Marseille
  - Almirall Investigational Sites#1, Marseille
  - Almirall Investigational Sites#6, Montpellier
  - Almirall Investigational Sites#4, Toulouse
- Germany (17):
  - Almirall Investigational Sites#8, Berlin
  - Almirall Investigational Sites#9, Berlin
  - Almirall Investigational Sites#6, Berlin
  - Almirall Investigational Sites#14, Berlin
  - Almirall Investigational Site#7, Berlin
  - Almirall Investigational Sites#12, Bonn
  - Almirall Investigational Sites#10, Cologne
  - Almirall Investigational Sites#3, Dortmund
  - Almirall Investigational Sites#13, Frankfurt
  - Almirall Investigational Sites#15, Gelsenkirchen
  - Almirall Investigational Sites#1, Großhansdorf
  - Almirall Investigational Sites#5, Hamburg
  - Almirall Investigational Sites#4, Hamburg
  - Almirall Investigational Site#16, Hanover
  - Almirall Investigational Sites#18, Jena
  - Almirall Investigational Sites#11, Mainz
  - Almirall Investigational Site#2, Rüdersdorf
- Hungary (13):
  - Almirall Investigational Sites#13, Budapest
  - Almirall Investigational Sites#4, Budapest
  - Almirall Investigational Sites#1, Budapest
  - Almirall Investigational Sites#2, Budapest
  - Almirall Investigational Sites#6, Debrecen
  - Almirall Investigational Sites#5, Debrecen
  - Almirall Investigational Sites#7, Deszk
  - Almirall Investigational Sites#10, Dunaüjváros
  - Almirall Investigational Sites#9, Mátraháza
  - Almirall Investigational Sites#12, Pécs
  - Almirall Investigational Sites#11, Ráckeve
  - Almirall Investigational Sites#3, Százhalombatta
  - Almirall Investigational Sites#8, Zalaegerszeg
- Italy (3):
  - Almirall Investigational Sites#3, Cagliari
  - Almirall Investigational Sites#1, Genova
  - Almirall Investigational Sites#10, Pisa
- Almirall Investigational Sites#8, Cusco, Peru
- Poland (22):
  - Almirall Investigational Sites#12, Bialystok
  - Almirall Investigational Sites#9, Bialystok
  - Almirall Investigational Sites#19, Elblag
  - Almirall Investigational Sites#18, Gdansk
  - Almirall Investigational Sites#20, Iława
  - Almirall Investigational Sites#7, Lodz
  - Almirall Investigational Sites#1, Lodz
  - Almirall Investigational Sites#8, Lublin
  - Almirall Investigational Sites#24, Olsztyn
  - Almirall Investigational Sites#5, Olsztyn
  - Almirall Investigational Sites#21, Poznan
  - Almirall Investigational Sites#16, Poznan
  - Almirall Investigational Site#11, Proszowice
  - Almirall Investigational Sites#2, Ruda Śląska
  - Almirall Investigational Sites#13, Rudka
  - Almirall Investigational Sites#4, Sopot
  - Almirall Investigational Sites#14, Szczecin
  - Almirall Investigational Sites#15, Tarnów
  - Almirall Investigational Sites#6, Tarnów
  - Almirall Investigational Sites#25, Warsaw
  - Almirall Investigational Sites#23, Wilkowice-Bystra
  - Almirall Investigational Site#10, Wroclaw
- Russia (11):
  - Almirall Investigational Sites#5, Kazan'
  - Almirall Investigational Sites#2, Moscow
  - Almirall Investigational Sites#14, Moscow
  - Almirall Investigational Sites#6, Moscow
  - Almirall Investigational Sites#13, Novosibirsk
  - Almirall Investigational Sites#10, Saint Petersburg
  - Almirall Investigational Sites#3, Saint Petersburg
  - Almirall Investigational Sites#4, Saint Petersburg
  - Almirall Investigational Sites#8, Tomsk
  - Almirall Investigational Sites#12, Tomsk
  - Almirall Investigational Sites#7, Yekaterinburg
- South Africa (13):
  - Almirall Investigational Sites#8, Bloemfontein
  - Almirall Investigational Sites#11, Bloemfontein
  - Almirall Investigational Sites#3, Bloemfontein
  - Almirall Investigational Sites#10, Cape Town
  - Almirall Investigational Sites#1, Cape Town
  - Almirall Investigational Sites#12, Cape Town
  - Almirall Investigational Sites#15, Cape Town
  - Almirall Investigational Sites#2, Durban
  - Almirall Investigational Sites#9, George
  - Almirall Investigational Sites#4, Port Elizabeth
  - Almirall Investigational Sites#5, Pretoria
  - Almirall Investigational Sites#14, Pretoria
  - Almirall Investigational Sites#6, Pretoria
- Spain (5):
  - Almirall Investigational Sites#6, Badalona
  - Almirall Investigational Sites#8, Barcelona
  - Almirall Investigational Sites#7, Barcelona
  - Almirall Investigational Sites#3, Madrid
  - Almirall Investigational Sites#5, Valencia
- Ukraine (6):
  - Almirall Investigational Sites#4, Donetsk
  - Almirall Investigational Sites#3, Kharkiv
  - Almirall Investigational Sites#1, Kyiv
  - Almirall Investigational Sites#2, Kyiv
  - Almirall Investigational Sites#7, Kyiv
  - Almirall Investigational Sites#5, Zaporizhzhya

REFERENCES:
- [Derived] McGarvey L, Morice AH, Smith JA, Birring SS, Chuecos F, Seoane B, Jarreta D. Effect of aclidinium bromide on cough and sputum symptoms in moderate-to-severe COPD in three phase III trials. BMJ Open Respir Res. 2016 Dec 8;3(1):e000148. doi: 10.1136/bmjresp-2016-000148. eCollection 2016. PMID 28074135
- [Derived] Jones PW, Leidy NK, Hareendran A, Lamarca R, Chuecos F, Garcia Gil E. The effect of aclidinium bromide on daily respiratory symptoms of COPD, measured using the Evaluating Respiratory Symptoms in COPD (E-RS: COPD) diary: pooled analysis of two 6-month Phase III studies. Respir Res. 2016 May 23;17(1):61. doi: 10.1186/s12931-016-0372-1. PMID 27215749
- [Derived] Jones PW, Lamarca R, Chuecos F, Singh D, Agusti A, Bateman ED, de Miquel G, Caracta C, Garcia Gil E. Characterisation and impact of reported and unreported exacerbations: results from ATTAIN. Eur Respir J. 2014 Nov;44(5):1156-65. doi: 10.1183/09031936.00038814. Epub 2014 Sep 18. PMID 25234803
- [Derived] Jones PW, Singh D, Bateman ED, Agusti A, Lamarca R, de Miquel G, Segarra R, Caracta C, Garcia Gil E. Efficacy and safety of twice-daily aclidinium bromide in COPD patients: the ATTAIN study. Eur Respir J. 2012 Oct;40(4):830-6. doi: 10.1183/09031936.00225511. Epub 2012 Mar 22. PMID 22441743
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 103 sites (100/103 randomised patients), 10 sites in the Czech Republic, 5 in France, 17 in Germany, 13 in Hungary, 3 in Italy, 1 in Peru, 21 in Poland, 10 in the Russian Federation, 5 in Spain, 13 in South Africa and 5 in the Ukraine. The first patient was screened in Oct 2009 and the last patient visit was in Nov 2010.
Pre-assignment Details: Patients fulfilling inclusion/exclusion criteria at the time of the Screening Visit were entered into a run-in period of 14±3 days to assess patient's disease stability.
Groups:
- Aclidinium Bromide 400 μg Bid: Aclidinium bromide 400 μg twice-daily via inhalation
- Placebo: Placebo via inhalation
Period: Overall Study
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Started | 277 (280 patients were randomized, but baseline data was missing from 3 patients in one center) | 269 (272 patients were randomized, but baseline data was missing from 3 patients in one center) | 273 (276 patients were randomized, but baseline data was missing from 3 patients in one center)
Completed | 253 | 252 | 232
Not Completed | 24 | 17 | 41
Not completed — Adverse Event | 8 | 4 | 6
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 7 | 17
Not completed — COPD exacerbation | 3 | 4 | 5
Not completed — Lack of Efficacy | 2 | 0 | 8
Not completed — Other | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo | Total
Number analyzed (Participants) | 277 | 269 | 273 | 819
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 169 | 161 | 179 | 509
  >=65 years | 108 | 108 | 94 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.8) | 62.9 (8.4) | 62.0 (8.0) | 62.4 (8.0)
Gender [Count of Participants; unit: Participants]
  Female | 96 | 87 | 84 | 267
  Male | 181 | 182 | 189 | 552
Region of Enrollment [Number; unit: participants]
  Spain | 6 | 7 | 5 | 18
  Ukraine | 8 | 8 | 11 | 27
  Russian Federation | 14 | 16 | 15 | 45
  Italy | 4 | 2 | 2 | 8
  France | 8 | 8 | 8 | 24
  Hungary | 35 | 30 | 32 | 97
  Czech Republic | 22 | 20 | 19 | 61
  Poland | 79 | 74 | 77 | 230
  South Africa | 46 | 47 | 48 | 141
  Germany | 55 | 57 | 56 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) Forced Expiratory Volume in the First Second (FEV1) at Week 24 on Treatment
Time Frame: Baseline and Week 24
Population: Intention-to-treat (ITT) population: all randomised patients who took at least one dose of Investigational Medicinal Product and who had a baseline and at least 1 post-baseline FEV1 assessment.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 277 | 269 | 273
Liters | 0.026 (0.016) | 0.055 (0.016) | -0.073 (0.016)

2. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) Forced Expiratory Volume in the First Second (FEV1) at Week 12 on Treatment
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 277 | 269 | 273
Liters | 0.030 (0.014) | 0.058 (0.015) | -0.047 (0.015)

3. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in the First Second (FEV1) at Week 24 on Treatment
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 277 | 269 | 273
Liters | 0.206 (0.017) | 0.231 (0.017) | 0.022 (0.017)

4. Secondary Outcome: Percentage of Patients Who Achieved at Least a 1-unit Decrease From Baseline in TDI Focal Score at Week 24 on Treatment
Description: Number of patients achieving a clinically meaningful improvement (≥1-unit) in Transition Dyspnoea Index (TDI) focal score at Week 24 on Treatment
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 270 | 262 | 257
Percentage of participants
  Yes (% Patients with a 1-unit decrease) | 53.3 | 56.9 | 45.5
  No (% Patients with a 1-unit decrease) | 46.7 | 43.1 | 54.5

5. Secondary Outcome: Percentage of Patients Who Achieved at Least a 4-unit Decrease From Baseline in the SGRQ Total Score at Week 24 on Treatment
Description: Number of patients who achieved a clinically meaningful improvement (≥4-units) in Saint George Respiratory Questionnaire (SGRQ) total score at week 24 on treatment
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Number analyzed (Participants) | 275 | 269 | 271
Percentage of participants
  Yes (% Patients with 4-unit decrease) | 56.0 | 57.3 | 41.0
  No (% Patients with 4-unit decrease) | 44.0 | 42.8 | 59.0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 12/277 | 15/269 | 15/273
Other Adverse Events (participants affected / at risk) | 44/277 | 38/269 | 56/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 200 μg Bid (N=277) | Aclidinium Bromide 400 μg Bid (N=269) | Placebo (N=273)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 10 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left vetricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ligament ruptures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortis stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian atery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Mixed deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 200 μg Bid (N=277) | Aclidinium Bromide 400 μg Bid (N=269) | Placebo (N=273)
Chronic obstructivce pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 44 | 38 | 56
Headache (Nervous system disorders) | 30 | 33 | 22
Nasopharyngitis (Infections and infestations) | 32 | 30 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.